CLINICAL TRIAL: NCT02994875
Title: Functional Magnetic Resonance Imaging of N-acetylcysteine in Cocaine Dependence
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1510016617; 1K01DA039299-01A1 (NIH)
Record Dates: First submitted 2016-07-11; First posted 2016-12-16 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo First (Placebo Comparator): Placebo - Participants will receive placebo for one week. Following a two-week washout period, they will receive NAC for one week. NAC is an FDA-approved dietary supplement with antioxidant properties that is available over-the-counter. NAC has no contraindications
  Interventions: Other: Placebo
- NAC First (Active Comparator): N-acetylcysteine - Participants will receive NAC for one week. Following a two-week washout period, they will receive placebo for one week. NAC is an FDA-approved dietary supplement with antioxidant properties that is available over-the-counter. NAC has no contraindications
  Interventions: Dietary Supplement: N-acetylcysteine

INTERVENTIONS:
Dietary Supplement: N-acetylcysteine — NAC is an FDA-approved dietary supplement with antioxidant properties that is available over-the-counter. NAC has no contraindications.
  Other Names: NAC
  Arms: NAC First
Other: Placebo — Sugar pill
  Arms: Placebo First

SUMMARY:
The objective of this research is to identify the functional neural mechanisms (as assessed using fMRI) of short-term N-acetylcysteine (NAC) administration among methadone-maintained individuals with cocaine dependence.

DETAILED DESCRIPTION:
The objective of this research is to identify the functional neural mechanisms (as assessed using fMRI) of short-term N-acetylcysteine (NAC) administration among methadone-maintained individuals with cocaine dependence. Specifically, this application proposes to conduct a randomized, double-blind, placebo-controlled, cross-over pilot study to examine the effects of 7-day NAC administration (2400mg/day) on the neural networks engaged during response inhibition (Go/No-Go task) and affective (emotion-regulation task) processes among cocaine-dependent, methadone-maintained individuals (n=40; 20 per treatment-order condition).

ELIGIBILITY:
Inclusion Criteria:

1. enrollment in the APT methadone program and maintained on a stable dose of methadone for ≥ 2 weeks
2. males or females, aged 18-65
3. confirmed DSM-IV diagnosis of current cocaine use disorder as assessed at the screening assessment
4. for women of a child-bearing age, acceptable birth control method
5. ability to commit to 4 weeks of study participation plus 1-month follow-up
6. willingness to be randomized to NAC or placebo
7. eligibility for MRI scanning and willingness to participate in MRI scanning.

Exclusion Criteria:

1. Do not meet DSM-IV criteria for cocaine-use disorder.
2. Meet DSM-IV psychiatric classifications for lifetime schizophrenia or bipolar disorder, or exhibit significant current suicidal or homicidal plans and intent such that hospitalization is required.
3. Meet DSM-IV criteria for current alcohol or other substance-use disorder dependence (with the exceptions of nicotine, cocaine and opioids).
4. Have previously taken or currently take NAC.
5. Have asthma (due to possible complications with NAC).
6. Cannot commit to 4-weeks of study participation or are unwilling to accept randomization.
7. Have any contraindications for MRI scanning (e.g., pregnancy, color-blindness, claustrophobia, metal implants that could interfere with MRI, any other contraindication to scanning).
8. Have lab work (complete blood count, urinalysis, liver function tests, thyroid function tests) suggesting the presence of any abnormalities or have a significant or unstable medical illness.
9. Are women who are pregnant or of a child-bearing age who do not agree to adequate contraception to prevent pregnancy during the study period.
10. Are not fluent in English.
11. Do not have at least a 6th grade reading level.
12. Cannot provide written, informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Change in neural network engagement measured using functional magnetic resonance imaging | 4 weeks
  The primary outcome measure for this study is change (NAC versus placebo) in neural network engagement during fMRI task performance.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Yip, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided